CLINICAL TRIAL: NCT05377645
Title: The Effects of Cervical Mobilization on Cognitive Performance and Anxiety in Individuals With Non-Specific Neck Pain
Brief Title: The Effects of Cervical Mobilization on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İSMAİL CEYLAN (Other)
Responsible Party: Sponsor-Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12068451747
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Pain, Chronic
Keywords: Pain Mobilisation; Anxiety
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical mobilization (Experimental): Mobilization Cyriax's cervical mobilization technique and traditional physiotherapy were applied to the intervention group. For Cyriax Mobilization technique, the patient was asked to lying supine position. Cervical ROM applied all directions. Also AP and ML glides applied to the cervical region. The treatment was done 3 times a week for 2 weeks. Also traditional physiotherapy techniques were applied to the experimental group. Traditional physiotherapy techniques were applied to the intervention group. Conventional TENS type was used. Continuous ultrasound type was applied with full contact technique.. And; isometric cervical strengthening exercises applied. The treatment was done 3 times a week for 2 weeks.
  Interventions: Other: Cyriax mobilization + traditional physiotherapy
- Traditional physiotherapy (Active Comparator): Traditional physiotherapy techniques were applied to the intervention group. Conventional TENS type was used. Current transition time was set as 50-100 µs. TENS application is performed at a frequency of 100 Hertz for 20 minutes in amplitude that does not cause muscle contraction in the patient and creates a feeling of numbness and tingling. Continuous ultrasound type was applied with full contact technique. Ultrasound treatment was applied over the suboccipital area with circular movements towards the proximal and distal at a speed of 1-2.5 cm per second, at a dose of 1 W / cm2, for 6 minutes, with a frequency of 3 MHz. And; isometric cervical strengthening exercises applied. The treatment was done 3 times a week for 2 weeks.
  Interventions: Other: Cyriax mobilization + traditional physiotherapy

INTERVENTIONS:
Other: Cyriax mobilization + traditional physiotherapy — TENS, US, exercise

SUMMARY:
Non spesific cervical pain syndromes are the most common cervical pathologies encountered in clinical practice. Non spesific cervical pain syndrome occurs as a result of postural deformities.

Massage and mobilization techniques are used in the treatment of Non spesific cervical pain syndrome due to their analgesic effects. The Cyriax mobilization technique is a manual therapy method applies to correct the limitation of movement in the joint and to relieve pain and functional disorders. Many studies have shown that Cyriax mobilization technique provides faster and momentary painless joint movement compared to other physical therapy modalities. Cervical mobilisation techniques also have regulator effect on autonomic nerve system. Cervical mobilisation also has positive effects on anxiety and tension.

DETAILED DESCRIPTION:
In this study, 32 patients with age range 18-65 who applied to Kırşehir Ahi Evran University Training and Research Hospital were examined. The individuals included in the study were divided into two groups according to the paired randomization method. These groups were control and intervention groups. Traditional physiotherapy methods were applied to the control group, traditional physiotherapy and Cyriax mobilisation techniques were applied to the intervention group. Traditional physiotherapy methods were included; Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US), isometric strengthening exercises.

For the evaluation of patients; Visual Analogue Scale (VAS), cervical goniometric measurements, Lowett muscle test, Burdon Test and Beck Anxiety Test were used.

ELIGIBILITY:
Inclusion Criteria:

* Who had cervical pain longer than six weeks
* Getting at least five points from Neck Disability Index

Exclusion Criteria:

* Who had neck surgery,
* Who had traumatic spinal cord injury,
* Clinical diagnosis of radiculopathy,
* Clinical diagnosis of myelopathy (sensory or motor deficit),
* Clinical diagnosis of neurological or rheumatologic disease and structural scoliosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 0-2 weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, İç Anadolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calixtre LB, Oliveira AB, de Sena Rosa LR, Armijo-Olivo S, Visscher CM, Alburquerque-Sendin F. Effectiveness of mobilisation of the upper cervical region and craniocervical flexor training on orofacial pain, mandibular function and headache in women with TMD. A randomised, controlled trial. J Oral Rehabil. 2019 Feb;46(2):109-119. doi: 10.1111/joor.12733. Epub 2018 Oct 26. PMID 30307636